CLINICAL TRIAL: NCT00820469
Title: Influence of Plasma Exchange Therapy on the Pharmacokinetics of Rituximab in Patients Treated for Autoimmune Disorders.
Brief Title: Study of the Influence of Plasma Exchange on the Pharmacokinetics of Rituximab
Acronym: PK-rituximab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 07 140 03
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Renal Transplant; Autoimmune Diseases
Keywords: Rituximab; Plasma exchange; Autoimmune diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients treated by rituximab
  Interventions: Drug: Rituximab 375
- 2 (Experimental): Patients treated by rituximab and plasma exchange
  Interventions: Drug: rituximab 1000

INTERVENTIONS:
Drug: Rituximab 375 — rituximab 375 mg/m2 IV weekly, during 4 weeks
  Arms: 1
Drug: rituximab 1000 — rituximab 1000 mg IV, two infusions on day 1 and day 15
  Arms: 2

SUMMARY:
Rituximab (a monoclonal antibody raised against CD20) is used to treat various immune disorders. In some cases such as treatment of humoral acute rejection of renal transplant, thrombotic thrombocytopenic purpura, vasculitis or cryoglobulinemia, rituximab is often associated with plasma exchange. The pharmacokinetic of the rituximab can be affected by plasma exchange but the knowledge is poor in this matter.

The aim of the study is to explore the influence of plasma exchange on the pharmacokinetic of rituximab.

The results of this study should conclude if plasma exchange leads to a significant decrease of plasma concentration of rituximab or not, and if the decreased of the concentration is associated with a decrease in efficacy.

DETAILED DESCRIPTION:
Twenty patients will be enrolled: ten patients treated by rituximab and ten patients treated by rituximab and plasma exchange. The plasma concentration of rituximab and the efficacy of the treatment will be compared between the two groups of patients.

The enrollment in the study will not change the treatment of patients except for blood sampling.

Each patient will undergo fifteen blood samples between the start of infusion of rituximab and three months after the start of infusion. For the patients who will undergo plasma exchange, three additional blood samples will be performed at each plasma exchange (at the start, at the end and one day after the plasma exchange) and a sample of the plasma exchanged will be keep.

The plasma concentration of rituximab will be determined by ELISA method (Enzyme Linked ImmunoSorbent Assay) The pharmacokinetic analyse will consist in the determination of the Area Under the Concentration Curve (AUC) by a non compartmental approach.

The AUC levels will be compared (using the t Student test) between the two populations of patients (patients treated by rituximab, versus patients treated by rituximab and plasma exchange) The efficacy of the treatment will be evaluated by the CD19+ B Cell count.

ELIGIBILITY:
Inclusion Criteria:

* Patient who should be treated by rituximab for various autoimmune diseases or humoral acute rejection of renal transplant
* Patient older than 18 years old
* Patient who have signed the written informed consent form

Exclusion Criteria:

* Patient presenting a contra indication to rituximab (hypersensitivity, active infection, severe cardiac failure (NYHA class IV))
* Blood sampling impossibility
* Pregnant or breasting women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the total AUC levels between 2 arms : patients treated by rituximab alone or patients treated by rituximab and plasma exchange | Determination on the overall plasma concentration profile between the start of infusion and three months after the start of infusion

SECONDARY OUTCOMES:
Determination of amount rituximab eliminated during a plasma exchange | At each plasma exchange
Evaluation of the efficacy of the treatment by CD19+B Cell count | 15 dyas, 1, 2, 3, 6 and 9 months after rituximab infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Pourrat, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

REFERENCES:
- [Result] Puisset F, White-Koning M, Kamar N, Huart A, Haberer F, Blasco H, Le Guellec C, Lafont T, Grand A, Rostaing L, Chatelut E, Pourrat J. Population pharmacokinetics of rituximab with or without plasmapheresis in kidney patients with antibody-mediated disease. Br J Clin Pharmacol. 2013 Nov;76(5):734-40. doi: 10.1111/bcp.12098. PMID 23432476